CLINICAL TRIAL: NCT02155335
Title: Preference for a Prefilled Syringe or Smartject™ Device for Delivering SIMPONI (Golimumab) in Patients Suffering From Moderate to Severe Ulcerative Colitis
Brief Title: Preference for a Prefilled Syringe or Smartject™ Device for Delivering Golimumab in Participants Suffering From Moderate-to-severe Ulcerative Colitis (MK-8259-027)
Acronym: SMART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 8259-027; 2014-000656-29 (EudraCT Number)
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prefilled Syringe→Smartject™ Device (Experimental): Golimumab 50 mg supplied in a prefilled syringe administered 2 times (once by the treating physician and then by the participant under the supervision of the treating physician). Participant is then administered Golimumab 50 mg supplied in the Smartject 2 times, first by the physician and then by the participant. Participants receive a total of 200 mg of golimumbab).
  Interventions: Drug: Prefilled Syringe delivery of Golimumab
- Smartject™ Device→ Prefilled Syringe (Experimental): Golimumab 50 mg supplied in a Smartject administered 2 times (once by the treating physician and then by the participant under the supervision of the treating physician). Participant is then administered Golimumab 50 mg supplied a prefilled syringe 2 times, first by the physician and then by the participant. Participants receive a total of 200 mg of golimumbab.
  Interventions: Drug: Smartject Device delivery of Golimumab

INTERVENTIONS:
Drug: Prefilled Syringe delivery of Golimumab — Golimumab 50 mg solution for subcutaneous injection using prefilled syringe
  Arms: Prefilled Syringe→Smartject™ Device
Drug: Smartject Device delivery of Golimumab — Golimumab 50 mg solution for subcutaneous injection using Smartject Device.
  Arms: Smartject™ Device→ Prefilled Syringe

SUMMARY:
This study is designed to determine whether ulcerative colitis participants prefer delivery of golimumab via a prefilled syringe or the Smartject™ device.

ELIGIBILITY:
Inclusion Criteria:

* Anti-tumor necrosis factor (anti-TNF) naive participants with a diagnosis of moderate-to-severe ulcerative colitis.
* Mayo clinic score >= 6, including endoscopic subscore >=2;
* Previous conventional therapy for a period of at least 3 months with aminosalicylates and at least 3 months with corticosteroids or 6-mercaptopurine (6-MP) or azathioprine (AZA), unless the participant is intolerant to, or has contraindications to these treatments;
* Anti-TNF experienced participants with an established diagnosis of moderate-to-severe ulcerative colitis, either not responding or partially responding to treatment with Remicade (infliximab). The participant must also meet the following criteria prior to initiating first-line anti-TNF treatment: Mayo score ≥ 6, including an endoscopic subscore ≥ 2; and previous conventional therapy of at least 3 months with aminosalicylates and at least 3 months with corticosteroids or 6-mercaptopurine (6-MP) or azathioprine (AZA), unless the participant is intolerant to or have medical contraindications for such therapies (should be documented);
* Sexually active women of child-bearing potential must agree to use a medically accepted method of contraception while receiving study drug and for 6 months after the stop of study drug

Exclusion Criteria:

* Has a history of prior self-injection for any reason;
* Has concomitant use of other biologic agents;
* Has active tuberculosis (TB) within 12 months prior to the first injection or has suspected latent TB as indicated by a positive tuberculin skin test.
* Has an active clinical non-tuberculous mycobacterial infection or opportunistic infection within 6 months prior to the first injection;
* Has had an active infection and/or serious infection within 6 months prior to the first study drug administration;
* Has had a live viral or bacterial vaccination within 3 months prior to the first study injection or Bacillus Calmette-Guerin vaccination within 12 months prior to the first study drug injection;
* Has evidence of heart failure of New York Heart Association class 3-4;
* Has a history of demyelinating disease such as multiple sclerosis or optic neuritis;
* Has a history of systemic lupus erythematosus;
* Has a history of lymphoproliferative disease, or any unknown malignancy or history of malignancy within the prior 5 years, with the exception of non-melanoma skin cancer that has been treated with no evidence of recurrence;
* Has had an active hepatitis B infection;
* Has an allergy or sensitivity to golimumab or its excipients;
* Is pregnant or breast feeding;
* Is sensitive to latex.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2015-10-05 (Actual); Study Completion 2015-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Bossuyt P, Baert F, D'Heygere F, Nakad A, Reenaers C, Fontaine F, Franchimont D, Dewit O, Van Hootegem P, Vanden Branden S, Lambrecht G, Ferrante M; Belgian IBD Research and Development Group. Early Mucosal Healing Predicts Favorable Outcomes in Patients With Moderate to Severe Ulcerative Colitis Treated With Golimumab: Data From the Real-life BE-SMART Cohort. Inflamm Bowel Dis. 2019 Jan 1;25(1):156-162. doi: 10.1093/ibd/izy219. PMID 29920582

RESULTS

PARTICIPANT FLOW:
Groups:
- Prefilled Syringe→Smartject™ Device: Golimumab 50 mg supplied in a prefilled syringe administered 2 times (once by the treating physician and then by the participant under the supervision of the treating physician). Participant than is administered Golimumab 50 mg supplied in the Smartject 2 times, first by the physician and then by the participant. Participants receive a total of 200 mg of golimumbab.
- Smartject™ Device→ Prefilled Syringe: Golimumab 50 mg supplied in a Smartject administered 2 times (once by the treating physician and then by the participant under the supervision of the treating physician). Participant than is administered Golimumab 50 mg supplied a prefilled syringe 2 times, first by the physician and then by the participant. Participants receive a total of 200 mg of golimumbab.
Period: Period 1
Arm/Group | Prefilled Syringe→Smartject™ Device | Smartject™ Device→ Prefilled Syringe
Started | 50 | 50
Treated | 50 | 49
Completed | 50 | 49
Not Completed | 0 | 1
Period: Period 2
Arm/Group | Prefilled Syringe→Smartject™ Device | Smartject™ Device→ Prefilled Syringe
Started | 50 | 49
Completed | 50 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 1 enrolled participant withdrew prior to treatment.
Groups:
- All Treated Participants: All participants who received at least 1 injection from either prefilled syringe or Smartject
Arm/Group | All Treated Participants
Number analyzed (Participants) | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 57

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Prefer Prefilled Syringe, Smartject™ Device, or Are Undecided (Day of Injections)
Description: Golimumab 50 mg supplied in a prefilled syringe administered 2 times (once by the treating physician and then by the participant under the supervision of the treating physician). Participant is then administered Golimumab 50 mg supplied in the Smartject 2 times, first by the physician and then by the participant. Following the completion of the last injection, the participants completed a questionnaire in which they indicated if they preferred the syringe, the Smartject or were undecided as to which they preferred.
Time Frame: Day 0 (post last injection)
Population: All enrolled participants who met all inclusion and none of the exclusion criteria, received all four injections of golimumab according to the protocol, and completed the device preference questionnaire
Measure: Number; unit: Percentage of Participants
Groups:
- Per Protocl Set (PPS): All enrolled participants who met all inclusion and none of the exclusion criteria, received all four injections of golimumab according to the protocol, and completed the device preference questionnaire.
Arm/Group | Per Protocl Set (PPS)
Number analyzed (Participants) | 91
Percentage of Participants
  Preferred Prefilled Syringe | 20.9
  Preferred Smatject Device | 76.9
  Undecided | 2.2

2. Primary Outcome: Percentage of Participants Who Prefer Prefilled Syringe, Smartject™ Device, or Are Undecided (2 Weeks Post Injections)
Description: Golimumab 50 mg supplied in a prefilled syringe administered 2 times (once by the treating physician and then by the participant under the supervision of the treating physician). Participant than is administered Golimumab 50 mg supplied in the Smartject 2 times, first by the physician and then by the participant. Participants completed a questionnaire 2 weeks after the injections in which they indicated if they preferred the syringe, the Smartject or were undecided as to which they preferred.
Time Frame: Day 14 (2 weeks post injections)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Per Protocl Set (PPS)
Number analyzed (Participants) | 91
Percentage of Participants
  Preferred Prefilled Syringe | 26.4
  Preferred Smatject Device | 71.4
  Undecided | 2.2

ADVERSE EVENTS:
Time Frame: up to 14 days post injections
Description: The study was crossover using 2 types of injection methods per participant, without a wash-out period between injection types. It was not possible to relate an adverse event (AE) to a specific injection method. Hence, per protocol, AEs were summarized for all participants who received at least 1 dose of golimumab, regardless of injection type.
Arm/Group | All Treated Participants
Serious Adverse Events (participants affected / at risk) | 0/99
Other Adverse Events (participants affected / at risk) | 0/99

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the trial without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial.